CLINICAL TRIAL: NCT01086709
Title: Crossover Vaccination of Women Previously Randomized Into Protocol 04-C-N191(NCI)/IC-200403(INCIENSA)
Brief Title: Crossover Vaccination of Women Previously Randomized Into Protocol 04-C-N191
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910059; 10-C-N059
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-03-17

CONDITIONS: Cervical Neoplasia; HPV Infections
Keywords: Human Papillomavirus; Vaccine; Crossover; Hepatitis A; Hepatitis B
MeSH Terms: conditions — Papillomavirus Infections; Hepatitis A; Hepatitis B

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- National Cancer Institute Protocol 04-C-N191, also known as the Costa Rica Vaccine Trial, was a double-blind controlled study of the effectiveness of an experimental human papillomavirus (HPV) vaccine in preventing cervical cancer in young women in Costa Rica. Costa Rica was part of the first large study to show the association between HPV and cervical cancer, and the study contributed greatly to the understanding of this association. The women who have participated in the vaccine trial in Costa Rica are reaching the end of the follow-up period offered in the vaccine trial protocol, and as a result they are being offered the chance to have complementary vaccinations against HPV, hepatitis A, and hepatitis B.

Objectives:

* To offer participants in the Costa Rica Vaccine Trial the vaccine that they did not receive during the masked portion of the trial (HPV vaccine or hepatitis A vaccine) and hepatitis B vaccination.
* To collect information about exposure to known and suspected risk factors for HPV infection and cervical cancer from women who are receiving vaccination against HPV at crossover.

Eligibility:

- Women who participated in National Cancer Institute Protocol 04-C-N191.

Design:

* All participants will be offered vaccination against hepatitis B.
* Women who received the hepatitis A vaccine during the trial will be offered vaccination against HPV.
* Women who received the HPV vaccine during the trial will be offered vaccination against hepatitis A.
* Appropriate vaccinations (including a combined hepatitis A and hepatitis B vaccine) will be available to reduce the number of injections that participants will be asked to receive.
* All vaccines will be given according to the manufacturer's specifications for appropriate length of time between vaccine doses.

DETAILED DESCRIPTION:
Since the mid 1980 s, the Division of Cancer Epidemiology and Genetics of the National Cancer Institute in collaboration with investigators in Costa Rica has conducted studies regarding cervical cancer and HPV infection. The first effort was a case control study where Costa Rica was one of the Latin American countries included, and it was the first large epidemiological study to show the association between HPV and cervical cancer. The second study, consisting of a 10,049 women population-based cohort, the Guanacaste cohort, was carried out from 1993 until 2004, and has greatly contributed to the understanding of the natural history of HPV infection and its relationship with precancerous cervical lesions.

The profound knowledge of the natural history of HPV infection and cervical neoplasia in Guanacaste, Costa Rica together with the promising results of the different HPV vaccine trials led the National Cancer Institute, in collaboration with investigators in Costa Rica, to launch a community-based randomized phase III clinical trial to evaluate the efficacy of a virus-like particle HPV vaccine (henceforth referred to as the Costa Rica Vaccine Trial (CVT)).

The main objectives of the Costa Rica Vaccine Trial were to evaluate the efficacy of the candidate vaccine to prevent persisting HPV-16/18 infections and related histopathologically confirmed CIN2+ lesions among the according to protocol subcohort and the overall population enrolled in the study. In contrast, the objectives of this protocol are aimed at offering beneficial complementary vaccination to women enrolled in the trial with an additional objective to collect biological specimens from women receiving the HPV-16/18 vaccine to complement the information obtained during the masked phase of the trial. As an additional objective, we propose to collect information regarding exposure to known and suspected risk factors for HPV infection and cervical cancer and biological specimens during this crossover phase that will complement those collected during the masked phase of the Costa Rica Vaccine Trial.

Collection of risk factor information and biological specimens during this crossover phase will be restricted to women receiving vaccination against HPV 16/18 at crossover. These samples will permit a more complete and comprehensive evaluation of the vaccine immunogenicity. Also, those specimens will allow for ancillary analyses and studies (e.g., natural history of HPV infection acquisition/clearance) and to assist ongoing efforts to evaluate the longer-term impact of HPV-16/18 vaccination.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to receive crossover vaccination, participants must fulfill all of the following inclusion criteria:

* Participation Status: Women previously randomized into the HPV-16/18 vaccine trial 04-C-N191, also known as the Costa Rica Vaccine Trial.
* Planned Residence: Residents of Guanacaste or Puntarenas Province or willingness to visit one of the study clinics for participation.
* Consent: Written informed consent obtained prior to enrollment into the crossover protocol.

EXCLUSION CRITERIA:

The following criteria will be checked for all potential participants at the time of enrollment. If any apply, the participant will not be included in the study.

* History of (a) allergic reaction (e.g., difficulty breathing) after receipt of any vaccine, (b) hypersensitivity to latex.
* History of vaccine related adverse events during the vaccination phase that, at the discretion of the investigators, preclude vaccination during the crossover phase.
* Are receiving vaccination with Cervarix , are sexually experienced and of childbearing potential (i.e., not surgically sterilized), and are unwilling to use an effective method of birth control for 30 days before vaccination until 60 days after the last Cervarix vaccination (approximately 9 months). Acceptable forms of birth control include abstinence, surgical sterilization, hormonal contraceptives (e.g., oral, injectable, implant, and patch), intrauterine devices, and diaphragm or condom.
* History of chronic condition that per attending doctor opinion precludes her from receiving vaccination (e.g., no proper treatment available or participant is unwilling to stay under proper treatment).
* The participant has a diagnosed autoimmune illness (per the specific requirement of the INCIENSA IRB).
* The vaccine or vaccines the participant is interested in receiving are contraindicated in her case.

Ages: 21 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5444 (Actual)
Dates: Start 2010-01-27; Study Completion 2015-03-17

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hildesheim, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Proyecto Epidemiologico Guanaste (PEG), San José, Costa Rica

REFERENCES:
- [Background] Reeves WC, Brinton LA, Garcia M, Brenes MM, Herrero R, Gaitan E, Tenorio F, de Britton RC, Rawls WE. Human papillomavirus infection and cervical cancer in Latin America. N Engl J Med. 1989 Jun 1;320(22):1437-41. doi: 10.1056/NEJM198906013202201. PMID 2541336
- [Background] Herrero R, Brinton LA, Reeves WC, Brenes MM, Tenorio F, de Britton RC, Gaitan E, Garcia M, Rawls WE. Invasive cervical cancer and smoking in Latin America. J Natl Cancer Inst. 1989 Feb 1;81(3):205-11. doi: 10.1093/jnci/81.3.205. PMID 2536087
- [Background] Herrero R, Schiffman MH, Bratti C, Hildesheim A, Balmaceda I, Sherman ME, Greenberg M, Cardenas F, Gomez V, Helgesen K, Morales J, Hutchinson M, Mango L, Alfaro M, Potischman NW, Wacholder S, Swanson C, Brinton LA. Design and methods of a population-based natural history study of cervical neoplasia in a rural province of Costa Rica: the Guanacaste Project. Rev Panam Salud Publica. 1997 May;1(5):362-75. doi: 10.1590/s1020-49891997000500005. PMID 9180057
- [Derived] Panagiotou OA, Befano BL, Gonzalez P, Rodriguez AC, Herrero R, Schiller JT, Kreimer AR, Schiffman M, Hildesheim A, Wilcox AJ, Wacholder S; Costa Rica HPV Vaccine Trial (CVT) Group (see end of manuscript for full list of investigators). Effect of bivalent human papillomavirus vaccination on pregnancy outcomes: long term observational follow-up in the Costa Rica HPV Vaccine Trial. BMJ. 2015 Sep 7;351:h4358. doi: 10.1136/bmj.h4358. PMID 26346155